CLINICAL TRIAL: NCT00477581
Title: A Randomized, Double-Blind, Crossover Study to Compare the Effects of Exenatide and Sitagliptin on Postprandial Glucose in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Compare the Effects of Exenatide and Sitagliptin on Postprandial Glucose in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BCA403
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; sitagliptin; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: exenatide; Drug: sitagliptin
- Sequence B (Experimental)
  Interventions: Drug: exenatide; Drug: sitagliptin

INTERVENTIONS:
Drug: exenatide — subcutaneous injection (5mcg or 10mcg), twice a day
  Other Names: Byetta
Drug: sitagliptin — oral administration (100mg), once a day in the morning
  Other Names: Januvia

SUMMARY:
This purpose of this study is to compare the effect of exenatide to that of sitagliptin on 2-hour postprandial glucose in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with metformin for at least 2 months
* Has HbA1c 7.0% to 11.0%, inclusive, at screening
* Body mass index (BMI)25 kg/m^2 to 45 kg/m^2, inclusive
* List of medications that are not allowed or the patient has been on stable treatment for at least 2 months:

  * Hormone replacement therapy (female subjects)
  * Oral contraceptives (female subjects)
  * Antihypertensive agents
  * Lipid-lowering agents
  * Thyroid replacement therapy

Exclusion Criteria

* Has been treated with exenatide (BYETTA®) or any DPP-4 inhibitor prior to screening
* Received any study medication or participated in any type of clinical trial within 30 days prior to screening
* Has donated blood within 60 days of screening visit or is planning to donate blood during the study
* Treated with any of the following medications:

  * Sulfonylurea or Thiazolidinedione within 3 months of screening;
  * Alpha-glucosidase inhibitor, meglitinide, nateglinide, or pramlintide (SYMLIN®)within 30 days of screening;
  * Insulin within 2 weeks prior to screening or insulin for longer than 1 week within 6 months of screening;
  * Drugs that directly affect gastrointestinal motility, including but not limited to, anticholinergics, macrolide antibiotics, dopamine antagonists, opioids, and Reglan®(metoclopramide);
  * Systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR®) steroids known to have a high rate of systemic absorption;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Effect of Exenatide on postprandial glucose | 28 days
  To compare the effect of exenatide to that of sitagliptin on 2-hour postprandial glucose in subjects with type 2 diabetes mellitus

SECONDARY OUTCOMES:
Assessment of effect of exenatide to the effect of sitagliptin the acetaminophen absorption test, and 6-point self-monitored blood glucose (SMBG) profiles | 28 days
  To compare the effect of exenatide to the effect of sitagliptin on the following endpoints in subjects with type 2 diabetes mellitus: postprandial glucose, insulin, insulin secretion rate, glucagon, and triglycerides; gastric emptying, as assessed by the acetaminophen absorption test, and 6-point self-monitored blood glucose (SMBG) profiles

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (18):
- United States (18):
  - Research Site, Los Angeles, California
  - Research Site, Spring Valley, California
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, Butte, Montana
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] DeFronzo RA, Okerson T, Viswanathan P, Guan X, Holcombe JH, MacConell L. Effects of exenatide versus sitagliptin on postprandial glucose, insulin and glucagon secretion, gastric emptying, and caloric intake: a randomized, cross-over study. Curr Med Res Opin. 2008 Oct;24(10):2943-52. doi: 10.1185/03007990802418851. Epub 2008 Sep 10. PMID 18786299